CLINICAL TRIAL: NCT02676245
Title: Parent Education and Choice About Newborn Screening and Bloodspot Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Case Western Reserve University (Other); Intermountain Health Care, Inc. (Other); Albert Einstein College of Medicine (Other); University of California, San Francisco (Other); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Botkin, Professor of Pediatrics, Chief Division of Medical Ethics and Humanities, Associate Vice President for Research, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB_00060088; R01HG006266 (NIH)
Record Dates: First submitted 2015-11-17; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Neonatal Screening
Keywords: Prenatal Education; Residual Specimens

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Viewing NBS + DBS Educational Movies (Experimental): Group A: pregnant women who will view the NBS and residual specimen movies and printed materials during one visit between 30 and 40 weeks gestation.
  Interventions: Behavioral: Viewing Newborn Screening movie; Behavioral: Viewing Residual Dried Blood Spot movie
- Viewing NBS Educational Movie only (Experimental): Group B: pregnant women who will view the NBS movie only and printed materials at one visit between 30 and 40 weeks. The movies will be presented on a tablet PC.
  Interventions: Behavioral: Viewing Newborn Screening movie
- No Educational Interventions (No Intervention): Control Group: pregnant women who will receive no experimental intervention during pregnancy or the postpartum period but will receive whatever information is routinely provided by their OB clinic and/or delivery center.

INTERVENTIONS:
Behavioral: Viewing Newborn Screening movie — NBS Movie and printed brochure were viewed by the participants
  Arms: Viewing NBS + DBS Educational Movies; Viewing NBS Educational Movie only
Behavioral: Viewing Residual Dried Blood Spot movie — DBS Movie and and printed brochure were viewed by the participants
  Arms: Viewing NBS + DBS Educational Movies

SUMMARY:
To address the content, timing, efficacy, and impact of prenatal education about newborn screening generally and sample retention specifically.

DETAILED DESCRIPTION:
It is widely recognized that new parents receive insufficient information about newborn screening (NBS) and little or no information regarding the retention of residual newborn screening samples. Our current research (R01 HD058854) clearly demonstrates that parents are supportive of NBS and the research use of residual specimens, but they want information before the child is born and want an informed choice regarding the retention and use of residual samples. Previous research has outlined the basic elements of what parents want to know about NBS generally. However, given that many states are adopting an "opt-out" approach for residual samples, it is unclear what basic information parents want to know to enable an informed choice about this practice. While it is recognized that retention and use of residual NBS samples is a valuable research resource, there are prevalent concerns in the NBS community that discussion of this will lead some parents to decline NBS altogether. Some authorities have suggested that discussions of NBS and residual sample retention be conducted separately to reduce the risk that parents will confuse the issues and decline NBS altogether.

To address this the project has the following specific aims:

Specific Aim 1) To determine what pregnant women, young mothers, and their partners want to know regarding the retention and use of residual bloodspot samples

Specific Aim 2) To create multimedia educational tools to be used in the prenatal care environment that will provide basic information about NBS and the core information determined through Specific Aim 1 about residual sample retention and use.

Specific Aim 3) To determine the impact of the prenatal education intervention on parental knowledge, attitudes, and decisions regarding NBS services and the retention and use of residual samples in diverse populations of English and Spanish speaking pregnant women.

Specific Aim 4) To examine the normative/ethical implications of the results of SA3 for the conduct of state NBS programs. Recommendations on the content and timing of parental NBS education will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years) women
* Uncomplicated pregnancy
* English and Spanish speaking
* Partners of pregnant women who have give birth.

Exclusion Criteria:

* Women younger than 18 years
* Complicated pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Factual knowledge about newborn screening as assessed through a survey instrument designed for the project | 2-4 weeks after due date
  Knowledge of key items about newborn screening that were conveyed in the educational interventions
Factual knowledge about newborn blood spots retention and use as assessed through a survey instrument designed for the project | 2-4 weeks after due date
  Knowledge of key items about newborn dried blood spots that were conveyed in the educational interventions

SECONDARY OUTCOMES:
Knowledge of partners of the pregnant women regarding newborn screening based on a survey instrument designed for the study | 2-4 weeks after due date
  Knowledge of newborn screening
Knowledge of partners of the pregnant women regarding newborn dried blood spots retention and use based on a survey instrument designed for the study | 2-4 weeks after due date
  Knowledge of newborn dried blood spots
An attitude assessment regarding support for newborn screening programs | 2-4 weeks after due date
  Attitudes regarding support for newborn screening
An attitude assessment regarding support for retention and use of newborn residual dried blood spots | 2-4 weeks after due date
  Attitudes regarding support for newborn dried blood spots
The clinical choices made by participants regarding participation in newborn screening | 2-4 weeks after due date
  Parents choice about newborn screening
The clinical choices made by participants regarding participation in the retention and use of dried blood spots | 2-4 weeks after due date
  Parents choice about dried bloodspot retention

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Botkin, MD, MPH, Principal Investigator — University of Utah

REFERENCES:
- [Result] Botkin JR, Rothwell E, Anderson RA, Goldenberg A, Kuppermann M, Dolan SM, Rose NC, Stark L. What parents want to know about the storage and use of residual newborn bloodspots. Am J Med Genet A. 2014 Nov;164A(11):2739-44. doi: 10.1002/ajmg.a.36694. Epub 2014 Aug 4. PMID 25131714
- [Derived] Botkin JR, Rothwell E, Anderson RA, Rose NC, Dolan SM, Kuppermann M, Stark LA, Goldenberg A, Wong B. Prenatal Education of Parents About Newborn Screening and Residual Dried Blood Spots: A Randomized Clinical Trial. JAMA Pediatr. 2016 Jun 1;170(6):543-9. doi: 10.1001/jamapediatrics.2015.4850. PMID 27043416